CLINICAL TRIAL: NCT01027845
Title: Immunogenicity, Safety and Reactogenicity of GlaxoSmithKline Biologicals' Pneumococcal Vaccine GSK1024850A Following Primary and Booster Vaccination of Healthy Japanese Children
Brief Title: Primary and Booster Vaccination Study With Pneumococcal Vaccine GSK1024850A in Healthy Japanese Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112640; 2011-003710-16 (EudraCT Number)
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Results first posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Infections, Streptococcal
Keywords: Pneumococcal disease; Immunogenicity; Booster vaccination; Pneumococcal vaccine; Primary vaccination; Safety
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections | interventions — PHiD-CV vaccine; Pentetic Acid

ARMS (2):
- 10Pn Group (Experimental): Healthy male or female subjects, between 90 and 118 days of age who received 3 doses of Synflorix (10Pn) vaccine, administered intramuscularly on alternating (left/right) sides of the anterolateral thigh and DPT "KAKETSUKEN" Syringe (DTPa) vaccine administered subcutaneously on alternating (left/right) sides of the distal one third of the upper arm. Both vaccines were administered at 3, 4, and 5 months of age, followed by a booster dose at 17-19 months of age.
  Interventions: Biological: Pneumococcal vaccine GSK1024850A; Biological: DTPa
- DTPa Group (Active Comparator): Healthy male or female subjects, between 90 and 118 days of age who received 3 doses of the DPT "KAKETSUKEN" Syringe (DTPa) vaccine, administered subcutaneously on alternating (left/right) sides of the distal one third of the upper arm at 3, 4, and 5 months of age, followed by a booster dose at 17-19 months of age.
  Interventions: Biological: DTPa

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK1024850A — Intramuscular injection, 4 doses
  Other Names: Synflorix
  Arms: 10Pn Group
Biological: DTPa — Subcutaneous injection, 4 doses
  Other Names: DPT "KAKETSUKEN" Syringe

SUMMARY:
This study will aim to evaluate the immunogenicity, safety and reactogenicity of GlaxoSmithKline Biologicals' 10-valent pneumococcal conjugate vaccine GSK1024850A when co-administered with Japanese DTPa vaccine as a 3-dose primary immunization course in healthy Japanese children at 3, 4 and 5 months of age and as a booster vaccination at 17-19 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator/co-investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR(s)) can and will comply with the requirements of the protocol.
* A male or female between, and including, 90 and 118 days of age (3 months) at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of 36 to 42 weeks inclusive.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccine(s), or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before the first dose of study vaccine(s) and ending on the last study visit, with the exception of Haemophilus influenzae type b vaccine, Hepatitis B Vaccine, Bacille Calmette-Guérin vaccine, Oral Polio Vaccine, Japanese encephalitis, measles and rubella, varicella, mumps, and flu vaccines.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Administration of any pneumococcal vaccine since birth except for the DTPa group for whom vaccination with a licensed pneumococcal vaccine by catch-up schedule will be allowed only if the 2 vaccine doses are administered between Study Visit 4 and 5, i.e. from the second blood sampling timepoint (Visit 4) onwards and up to 7 days before the booster dose of the DTPa vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of, or intercurrent diphtheria, tetanus, pertussis disease.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study vaccines.
* Major congenital defects or serious chronic illness.
* History of any seizures or progressive neurological disease.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Child in care.
* Acute disease and/or fever at the time of enrolment.

Ages: 90 Days to 118 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2009-12-08 (Actual); Primary Completion 2010-08-13 (Actual); Study Completion 2011-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- Japan (11):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=2812

REFERENCES:
- [Background] Iwata S, Kawamura N, Kuroki H, Tokoeda Y, Miyazu M, Iwai A, Oishi T, Sato T, Suyama A, Francois N, Shafi F, Ruiz-Guinazu J, Borys D. Immunogenicity and safety of the 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) co-administered with DTPa vaccine in Japanese children: A randomized, controlled study. Hum Vaccin Immunother. 2015;11(4):826-37. doi: 10.1080/21645515.2015.1012019. PMID 25830489
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 112640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 360 subjects were enrolled in the study. All subjects received at least one vaccination dose.
Groups:
- 10Pn Group: Healthy male or female subjects, between 90 and 118 days of age who received, during primary vaccination phase, 3 doses of Synflorix (10Pn) vaccine, administered intramuscularly on alternating (left/right) sides of the anterolateral thigh and DPT "KAKETSUKEN" Syringe (DTPa) vaccine administered subcutaneously on alternating (left/right) sides of the distal one third of the upper arm. Both vaccines were administered at 3, 4, and 5 months of age, followed by a booster dose at 17-19 months of age (booster vaccination phase).
- DTPa Group: Healthy male or female subjects, between 90 and 118 days of age, who received, during the primary vaccination phase, 3 doses of the DPT "KAKETSUKEN" Syringe (DTPa) vaccine, administered subcutaneously on alternating (left/right) sides of the distal one third of the upper arm at 3, 4, and 5 months of age, followed by a booster dose at 17-19 months of age (booster vaccination phase). Subjects from this group who also received at least one dose of Prevenar (PCV7): Pfizer's (formerly Wyeth Lederle) 7-valent pneumococcal conjugate vaccine, given before pre-booster blood sample (as optional treatment considered as standard of care), were assigned to the DTPa + Prevenar Group in the booster phase, and subjects who did not receive any dose of Prevenar before pre-booster blood sample were assigned to the DTPa-no Prevenar Group in the booster phase. Some booster phase analyses were only performed on subjects of both pooled sub-groups, renamed as DTPa booster Group, at the time of the analysis..
- DTPa + Prevenar Group: Healthy male or female subjects, between 90 and 118 days of age, who received, during the primary vaccination phase, 3 doses of the DPT "KAKETSUKEN" Syringe (DTPa) vaccine, administered subcutaneously on alternating (left/right) sides of the distal one third of the upper arm at 3, 4, and 5 months of age, followed by a booster dose at 17-19 months of age (booster vaccination phase). Those subjects received at least one dose of Prevenar (PCV7): Pfizer's (formerly Wyeth Lederle) 7-valent pneumococcal conjugate vaccine, given before pre-booster blood sample and considered optional treatment as standard of care.
- DTPa - no Prevenar Group: Healthy male or female subjects, between 90 and 118 days of age, who received, during the primary vaccination phase, 3 doses of the DPT "KAKETSUKEN" Syringe (DTPa) vaccine, administered subcutaneously on alternating (left/right) sides of the distal one third of the upper arm at 3, 4, and 5 months of age, followed by a booster dose at 17-19 months of age (booster vaccination phase). Those subjects did not receive any dose of Prevenar vaccination before pre-booster blood sample.
Period: Primary Vaccination Phase
Arm/Group | 10Pn Group | DTPa Group | DTPa + Prevenar Group | DTPa - no Prevenar Group
Started | 237 | 123 | 0 (Subjects were not yet assigned to this group at the time of the primary vaccination) | 0 (Subjects were not yet assigned to this group at the time of the primary vaccination)
Completed | 233 | 122 | 0 | 0
Not Completed | 4 | 1 | 0 | 0
Not completed — Serious Adverse Event | 2 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Migrated/moved from study area | 0 | 1 | 0 | 0
Period: Booster Vaccination Phase
Arm/Group | 10Pn Group | DTPa Group | DTPa + Prevenar Group | DTPa - no Prevenar Group
Started | 228 | 0 (Subjects from this group were assigned to DTPa+Prevenar&DTPa-No Prevenar Groups in the booster phase) | 119 | 1
Completed | 226 | 0 | 119 | 1
Not Completed | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Migrated/moved from study area | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10Pn Group | DTPa Group | Total
Number analyzed (Participants) | 237 | 123 | 360
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 13.6 (1.02) | 13.5 (1.1) | 13.57 (1.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 59 | 176
  Male | 120 | 64 | 184

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes (Primary Immunization)
Description: Concentrations were expressed as geometric mean concentrations (GMCs). Antibodies assessed for this outcome measure were those against the vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (ANTI-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F). The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 microgram per milliliter (µg/mL).
Time Frame: 1 month following primary immunization (at Month 3)
Population: The analysis was performed on the ATP cohort for immunogenicity for primary epoch, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after primary vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 10Pn Group | DTPa Group
Number analyzed (Participants) | 231 | 121
μg/mL
  Anti-1: number analyzed (Participants) | 231 | 119
  Anti-1 | 6.52 [5.85 to 7.26] | 0.04 [0.03 to 0.04]
  Anti-4: number analyzed (Participants) | 231 | 120
  Anti-4 | 6.54 [5.86 to 7.30] | 0.03 [0.03 to 0.03]
  Anti-5: number analyzed (Participants) | 231 | 119
  Anti-5 | 6.54 [5.94 to 7.21] | 0.05 [0.04 to 0.06]
  Anti-6B | 1.71 [1.43 to 2.05] | 0.03 [0.03 to 0.03]
  Anti-7F: number analyzed (Participants) | 231 | 120
  Anti-7F | 6.11 [5.50 to 6.78] | 0.03 [0.03 to 0.04]
  Anti-9V: number analyzed (Participants) | 231 | 119
  Anti-9V | 5.42 [4.81 to 6.10] | 0.03 [0.03 to 0.03]
  Anti-14: number analyzed (Participants) | 231 | 120
  Anti-14 | 10.03 [8.80 to 11.43] | 0.07 [0.06 to 0.09]
  Anti-18C | 16.59 [14.40 to 19.13] | 0.04 [0.03 to 0.04]
  Anti-19F: number analyzed (Participants) | 229 | 118
  Anti-19F | 17.39 [15.53 to 19.48] | 0.06 [0.05 to 0.07]
  Anti-23F: number analyzed (Participants) | 231 | 119
  Anti-23F | 2.17 [1.83 to 2.57] | 0.04 [0.03 to 0.04]
Statistical Analysis 1: Comparison: 10Pn Group; Immune response of Synflorix vaccine tested between subjects of the 10Pn Group of the study and healthy European subjects from the 10PN-PD-DIT-001 (105553) study (with following indication: 3-dose primary vaccination of infants between 6 to 12 weeks of age at the time of the first vaccination with Synflorix), that formed the 105553 10Pn Group. At 1 month after primary immunization (post-dose 3), ELISA GMC ratio (105553 10Pn Group over 10Pn Group) was calculated for pneumococcal serotype 1; Test type: Non-Inferiority — Comparability to the 105553 study in terms of non-inferiority was demonstrated if the upper limit (UL) of the two-sided 95% confidence interval(CI) on the GMC ratios (GMCs from 105553 10Pn Group over GMCs from 10Pn Group) were below a limit of 2-fold for all 10 vaccine pneumococcal serotypes. Number of participants analysed =1100 in the 105553 10Pn Group; GMC= 1.05 µg/mL with 95% CI = (1.00 to 1.10); GMC ratio = 0.16, 95% CI 2-sided [0.14 to 0.18]
Statistical Analysis 2: Comparison: 10Pn Group; Immune response of Synflorix vaccine tested between subjects of the 10Pn Group of the study and healthy European subjects from the 10PN-PD-DIT-001 (105553) study (with following indication: 3-dose primary vaccination of infants between 6 to 12 weeks of age at the time of the first vaccination with Synflorix), that formed the 105553 10Pn Group. At 1 month after primary immunization (post-dose 3), ELISA GMC ratio (105553 10Pn Group over 10Pn Group) was calculated for pneumococcal serotype 4; Test type: Non-Inferiority — Comparability to the 105553 study in terms of non-inferiority was demonstrated if the upper limit (UL) of the two-sided 95% confidence interval(CI) on the GMC ratios (GMCs from 105553 10Pn Group over GMCs from 10Pn Group) were below a limit of 2-fold for all 10 vaccine pneumococcal serotypes. Number of participants analysed =1106 in the 105553 10Pn Group; GMC= 1.45 µg/mL with 95% CI = (1.38 to 1.53); GMC ratio = 0.22, 95% CI 2-sided [0.2 to 0.25]
Statistical Analysis 3: Comparison: 10Pn Group; Immune response of Synflorix vaccine tested between subjects of the 10Pn Group of the study and healthy European subjects from the 10PN-PD-DIT-001 (105553) study (with following indication: 3-dose primary vaccination of infants between 6 to 12 weeks of age at the time of the first vaccination with Synflorix), that formed the 105553 10Pn Group. At 1 month after primary immunization (post-dose 3), ELISA GMC ratio (105553 10Pn Group over 10Pn Group) was calculated for pneumococcal serotype 5; Test type: Non-Inferiority — Comparability to the 105553 study in terms of non-inferiority was demonstrated if the upper limit (UL) of the two-sided 95% confidence interval(CI) on the GMC ratios (GMCs from 105553 10Pn Group over GMCs from 10Pn Group) were below a limit of 2-fold for all 10 vaccine pneumococcal serotypes. Number of participants analysed =1104 in the 105553 10Pn Group; GMC= 1.70 µg/mL with 95% CI = (1.62 to 1.78); GMC ratio = 0.26, 95% CI 2-sided [0.23 to 0.29]
Statistical Analysis 4: Comparison: 10Pn Group; Immune response of Synflorix vaccine tested between subjects of the 10Pn Group of the study and healthy European subjects from the 10PN-PD-DIT-001 (105553) study (with following indication: 3-dose primary vaccination of infants between 6 to 12 weeks of age at the time of the first vaccination with Synflorix), that formed the 105553 10Pn Group. At 1 month after primary immunization (post-dose 3), ELISA GMC ratio (105553 10Pn Group over 10Pn Group) was calculated for pneumococcal serotype 6B; Test type: Non-Inferiority — Comparability to the 105553 study in terms of non-inferiority was demonstrated if the upper limit (UL) of the two-sided 95% confidence interval(CI) on the GMC ratios (GMCs from 105553 10Pn Group over GMCs from 10Pn Group) were below a limit of 2-fold for all 10 vaccine pneumococcal serotypes. Number of participants analysed =1100 in the 105553 10Pn Group; GMC= 0.33 µg/mL with 95% CI = (0.30 to 0.36); GMC ratio = 0.19, 95% CI 2-sided [0.16 to 0.23]
Statistical Analysis 5: Comparison: 10Pn Group; Immune response of Synflorix vaccine tested between subjects of the 10Pn Group of the study and healthy European subjects from the 10PN-PD-DIT-001 (105553) study (with following indication: 3-dose primary vaccination of infants between 6 to 12 weeks of age at the time of the first vaccination with Synflorix), that formed the 105553 10Pn Group. At 1 month after primary immunization (post-dose 3), ELISA GMC ratio (105553 10Pn Group over 10Pn Group) was calculated for pneumococcal serotype 7F; Test type: Non-Inferiority — Comparability to the 105553 study in terms of non-inferiority was demonstrated if the upper limit (UL) of the two-sided 95% confidence interval(CI) on the GMC ratios (GMCs from 105553 10Pn Group over GMCs from 10Pn Group) were below a limit of 2-fold for all 10 vaccine pneumococcal serotypes. Number of participants analysed =1107 in the 105553 10Pn Group; GMC= 1.72 µg/mL with 95% CI = (1.64 to 1.80); GMC ratio = 0.28, 95% CI 2-sided [0.25 to 0.31]
Statistical Analysis 6: Comparison: 10Pn Group; Immune response of Synflorix vaccine tested between subjects of the 10Pn Group of the study and healthy European subjects from the 10PN-PD-DIT-001 (105553) study (with following indication: 3-dose primary vaccination of infants between 6 to 12 weeks of age at the time of the first vaccination with Synflorix), that formed the 105553 10Pn Group. At 1 month after primary immunization (post-dose 3), ELISA GMC ratio (105553 10Pn Group over 10Pn Group) was calculated for pneumococcal serotype 9V; Test type: Non-Inferiority — Comparability to the 105553 study in terms of non-inferiority was demonstrated if the upper limit (UL) of the two-sided 95% confidence interval(CI) on the GMC ratios (GMCs from 105553 10Pn Group over GMCs from 10Pn Group) were below a limit of 2-fold for all 10 vaccine pneumococcal serotypes. Number of participants analysed =1103 in the 105553 10Pn Group; GMC= 1.32 µg/mL with 95% CI = (1.25 to 1.38); GMC ratio = 0.24, 95% CI 2-sided [0.22 to 0.27]
Statistical Analysis 7: Comparison: 10Pn Group; Immune response of Synflorix vaccine tested between subjects of the 10Pn Group of the study and healthy European subjects from the 10PN-PD-DIT-001 (105553) study (with following indication: 3-dose primary vaccination of infants between 6 to 12 weeks of age at the time of the first vaccination with Synflorix), that formed the 105553 10Pn Group. At 1 month after primary immunization (post-dose 3), ELISA GMC ratio (105553 10Pn Group over 10Pn Group) was calculated for pneumococcal serotype 14; Test type: Non-Inferiority — Comparability to the 105553 study in terms of non-inferiority was demonstrated if the upper limit (UL) of the two-sided 95% confidence interval(CI) on the GMC ratios (GMCs from 105553 10Pn Group over GMCs from 10Pn Group) were below a limit of 2-fold for all 10 vaccine pneumococcal serotypes. Number of participants analysed =1100 in the 105553 10Pn Group; GMC= 2.90 µg/mL with 95% CI = (2.75 to 3.05); GMC ratio = 0.29, 95% CI 2-sided [0.25 to 0.33]
Statistical Analysis 8: Comparison: 10Pn Group; Immune response of Synflorix vaccine tested between subjects of the 10Pn Group of the study and healthy European subjects from the 10PN-PD-DIT-001 (105553) study (with following indication: 3-dose primary vaccination of infants between 6 to 12 weeks of age at the time of the first vaccination with Synflorix), that formed the 105553 10Pn Group. At 1 month after primary immunization (post-dose 3), ELISA GMC ratio (105553 10Pn Group over 10Pn Group) was calculated for pneumococcal serotype 18C; Test type: Non-Inferiority — Comparability to the 105553 study in terms of non-inferiority was demonstrated if the upper limit (UL) of the two-sided 95% confidence interval(CI) on the GMC ratios (GMCs from 105553 10Pn Group over GMCs from 10Pn Group) were below a limit of 2-fold for all 10 vaccine pneumococcal serotypes. Number of participants analysed =1102 in the 105553 10Pn Group; GMC= 1.66 µg/mL with 95% CI = (1.56 to 1.77); GMC ratio = 0.1, 95% CI 2-sided [0.09 to 0.12]
Statistical Analysis 9: Comparison: 10Pn Group; Immune response of Synflorix vaccine tested between subjects of the 10Pn Group of the study and healthy European subjects from the 10PN-PD-DIT-001 (105553) study (with following indication: 3-dose primary vaccination of infants between 6 to 12 weeks of age at the time of the first vaccination with Synflorix), that formed the 105553 10Pn Group. At 1 month after primary immunization (post-dose 3), ELISA GMC ratio (105553 10Pn Group over 10Pn Group) was calculated for pneumococcal serotype 19F; Test type: Non-Inferiority — Comparability to the 105553 study in terms of non-inferiority was demonstrated if the upper limit (UL) of the two-sided 95% confidence interval(CI) on the GMC ratios (GMCs from 105553 10Pn Group over GMCs from 10Pn Group) were below a limit of 2-fold for all 10 vaccine pneumococcal serotypes. Number of participants analysed =1104 in the 105553 10Pn Group; GMC= 1.84 µg/mL with 95% CI = (1.71 to 1.98); GMC ratio = 0.11, 95% CI 2-sided [0.09 to 0.12]
Statistical Analysis 10: Comparison: 10Pn Group; Immune response of Synflorix vaccine tested between subjects of the 10Pn Group of the study and healthy European subjects from the 10PN-PD-DIT-001 (105553) study (with following indication: 3-dose primary vaccination of infants between 6 to 12 weeks of age at the time of the first vaccination with Synflorix), that formed the 105553 10Pn Group. At 1 month after primary immunization (post-dose 3), ELISA GMC ratio (105553 10Pn Group over 10Pn Group) was calculated for pneumococcal serotype 23F; Test type: Non-Inferiority — Comparability to the 105553 study in terms of non-inferiority was demonstrated if the upper limit (UL) of the two-sided 95% confidence interval(CI) on the GMC ratios (GMCs from 105553 10Pn Group over GMCs from 10Pn Group) were below a limit of 2-fold for all 10 vaccine pneumococcal serotypes. Number of participants analysed =1102 in the 105553 10Pn Group; GMC= 0.53 µg/mL with 95% CI = (0.50 to 0.57); GMC ratio = 0.25, 95% CI 2-sided [0.21 to 0.29]

2. Secondary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes (Booster Immunization)
Description: Antibodies assessed for this outcome measure were those against the vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (ANTI-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F). Antibody concentrations were measured by 22F ELISA, expressed as GMCs, in μg/mL. The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 μg/mL. Antibody concentrations < 0.05 μg/mL were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
  Administration of catch-up pneumococcal vaccination with a licensed product other than Synflorix was allowed in the DTPa Group at least 7 days before DTPa vaccine booster dose. Thus, for this booster phase analysis, the DTPa Group was further split in DTPa + Prevenar Group and DTPa - no Prevenar Group.
Time Frame: Prior to (PRE, at Month 14-16 ) and one month after booster (POST, at Month 15-17) immunization
Population: The analysis was performed on the ATP cohort for immunogenicity for booster epoch, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component before and after booster vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 10Pn Group | DTPa + Prevenar Group | DTPa - no Prevenar Group
Number analyzed (Participants) | 216 | 114 | 1
μg/mL
  Anti-1 PRE: number analyzed (Participants) | 216 | 113 | 1
  Anti-1 PRE | 0.8 [0.69 to 0.92] | 0.04 [0.03 to 0.04] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-1 POST: number analyzed (Participants) | 214 | 114 | 1
  Anti-1 POST | 7.81 [6.91 to 8.82] | 0.04 [0.04 to 0.05] | 0.24 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-4 PRE: number analyzed (Participants) | 215 | 114 | 1
  Anti-4 PRE | 0.81 [0.7 to 0.93] | 0.85 [0.71 to 1.02] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-4 POST: number analyzed (Participants) | 213 | 114 | 1
  Anti-4 POST | 12.89 [11.41 to 14.56] | 0.78 [0.64 to 0.94] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-5 PRE | 1.22 [1.05 to 1.41] | 0.08 [0.07 to 0.1] | 0.05 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-5 POST: number analyzed (Participants) | 214 | 114 | 1
  Anti-5 POST | 8.81 [7.87 to 9.86] | 0.15 [0.12 to 0.17] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-6B PRE: number analyzed (Participants) | 215 | 114 | 1
  Anti-6B PRE | 0.93 [0.79 to 1.1] | 0.34 [0.27 to 0.44] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-6B POST: number analyzed (Participants) | 214 | 114 | 1
  Anti-6B POST | 3.66 [3.14 to 4.27] | 0.33 [0.25 to 0.42] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-7F PRE: number analyzed (Participants) | 215 | 114 | 1
  Anti-7F PRE | 1.48 [1.32 to 1.65] | 0.05 [0.04 to 0.05] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-7F POST: number analyzed (Participants) | 214 | 114 | 1
  Anti-7F POST | 10.68 [9.66 to 11.81] | 0.09 [0.08 to 0.11] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-9V PRE: number analyzed (Participants) | 212 | 114 | 1
  Anti-9V PRE | 1.81 [1.61 to 2.03] | 1.01 [0.83 to 1.25] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-9V POST: number analyzed (Participants) | 214 | 114 | 1
  Anti-9V POST | 12.79 [11.49 to 14.23] | 0.96 [0.79 to 1.17] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-14 PRE | 2.37 [2.04 to 2.74] | 3.17 [2.74 to 3.67] | 0.09 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-14 POST: number analyzed (Participants) | 214 | 114 | 1
  Anti-14 POST | 15.72 [13.97 to 17.69] | 2.92 [2.53 to 3.38] | 0.16 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-18C PRE | 2.18 [1.89 to 2.51] | 0.94 [0.79 to 1.11] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-18C POST: number analyzed (Participants) | 213 | 114 | 1
  Anti-18C POST | 34.9 [31.05 to 39.23] | 0.77 [0.65 to 0.92] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-19F PRE: number analyzed (Participants) | 215 | 114 | 1
  Anti-19F PRE | 2.92 [2.5 to 3.41] | 0.51 [0.38 to 0.68] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-19F POST: number analyzed (Participants) | 214 | 114 | 1
  Anti-19F POST | 28.72 [25.29 to 32.63] | 0.68 [0.51 to 0.91] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-23F PRE: number analyzed (Participants) | 213 | 114 | 1
  Anti-23F PRE | 1.14 [0.93 to 1.39] | 0.55 [0.42 to 0.73] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-23F POST: number analyzed (Participants) | 214 | 114 | 1
  Anti-23F POST | 7.68 [6.68 to 8.83] | 0.88 [0.7 to 1.12] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)

3. Secondary Outcome: Opsonophagocytic Titers Against Vaccine Pneumococcal Serotypes (Primary Immunization)
Description: Pneumococcal vaccine serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F and were calculated, expressed as geometric mean titers (GMTs). The seropositivity cut-off for the assay was ≥ 8. Antibody titers < 8 were given an arbitrary value of half the cut-off for the purpose of GMT calculation.
Time Frame: 1 month following primary immunization (at Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10Pn Group | DTPa Group
Number analyzed (Participants) | 224 | 116
Titers
  OPSONO-1: number analyzed (Participants) | 223 | 115
  OPSONO-1 | 619.8 [511.9 to 750.6] | 4.8 [4.2 to 5.5]
  OPSONO-4: number analyzed (Participants) | 221 | 115
  OPSONO-4 | 1184.6 [1043.7 to 1344.5] | 4.1 [3.9 to 4.3]
  OPSONO-5: number analyzed (Participants) | 224 | 115
  OPSONO-5 | 335.1 [286.4 to 392.1] | 4.2 [4 to 4.5]
  OPSONO-6B: number analyzed (Participants) | 222 | 116
  OPSONO-6B | 1926.6 [1559.6 to 2380] | 5 [4.2 to 5.9]
  OPSONO-7F: number analyzed (Participants) | 216 | 108
  OPSONO-7F | 7905.9 [6854.5 to 9118.6] | 69.5 [43.2 to 111.9]
  OPSONO-9V: number analyzed (Participants) | 219 | 108
  OPSONO-9V | 4063.4 [3565.8 to 4630.4] | 4.9 [4.2 to 5.6]
  OPSONO-14: number analyzed (Participants) | 217 | 103
  OPSONO-14 | 3392.4 [2962.5 to 3884.8] | 6.5 [5 to 8.5]
  OPSONO-18C: number analyzed (Participants) | 217 | 108
  OPSONO-18C | 893.2 [727.7 to 1096.2] | 4.8 [4 to 5.7]
  OPSONO-19F: number analyzed (Participants) | 219 | 115
  OPSONO-19F | 1254.6 [1031.1 to 1526.5] | 4.4 [4 to 4.9]
  OPSONO-23F: number analyzed (Participants) | 218 | 107
  OPSONO-23F | 4312.1 [3401.5 to 5466.5] | 6 [4.5 to 8]

4. Secondary Outcome: Opsonophagocytic Titers Against Vaccine Pneumococcal Serotypes (Booster Immunization)
Description: Pneumococcal vaccine serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F and were calculated, expressed as geometric mean titers (GMTs). The seropositivity cut-off for the assay was ≥ 8. Antibody titers < 8 were given an arbitrary value of half the cut-off for the purpose of GMT calculation. Administration of catch-up pneumococcal vaccination with a licensed product other than Synflorix was allowed in the DTPa Group at least 7 days before DTPa vaccine booster dose. Thus, for this booster phase analysis, the DTPa Group was further split in DTPa + Prevenar Group and DTPa - no Prevenar Group.
Time Frame: Prior to (PRE, at Month 14-16) and one month after booster (POST, at Month 15-17) immunization
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10Pn Group | DTPa + Prevenar Group | DTPa - no Prevenar Group
Number analyzed (Participants) | 214 | 113 | 1
Titers
  OPSONO-1 PRE | 45.9 [34.9 to 60.4] | 4.5 [4 to 5.1] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-1 POST: number analyzed (Participants) | 214 | 112 | 1
  OPSONO-1 POST | 2320.7 [1941.8 to 2773.6] | 4.7 [4.1 to 5.5] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-4 PRE: number analyzed (Participants) | 205 | 105 | 1
  OPSONO-4 PRE | 58.3 [43.6 to 77.9] | 79 [49.3 to 126.7] | 371 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-4 POST: number analyzed (Participants) | 214 | 109 | 1
  OPSONO-4 POST | 3863.1 [3319.7 to 4495.5] | 69.3 [43.1 to 111.5] | 493 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-5 PRE: number analyzed (Participants) | 212 | 113 | 1
  OPSONO-5 PRE | 22.9 [19.1 to 27.6] | 4.2 [3.9 to 4.5] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-5 POST: number analyzed (Participants) | 214 | 112 | 1
  OPSONO-5 POST | 686.7 [583.8 to 807.9] | 4.7 [4.1 to 5.3] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-6B PRE: number analyzed (Participants) | 212 | 110 | 1
  OPSONO-6B PRE | 191.2 [141.9 to 257.5] | 118.5 [66.3 to 211.7] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-6B POST: number analyzed (Participants) | 214 | 110 | 1
  OPSONO-6B POST | 1682.9 [1379.1 to 2053.7] | 119 [68.5 to 206.9] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-7F PRE: number analyzed (Participants) | 209 | 111 | 1
  OPSONO-7F PRE | 2244.8 [1921.9 to 2621.9] | 1014.7 [743.8 to 1384.1] | 588 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-7F POST: number analyzed (Participants) | 214 | 112 | 1
  OPSONO-7F POST | 14144.3 [12109.3 to 16521.4] | 1165.6 [855.7 to 1587.8] | 1278 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-9V PRE: number analyzed (Participants) | 213 | 113 | 1
  OPSONO-9V PRE | 520 [437.3 to 618.5] | 1081.6 [803.3 to 1456.4] | 4595 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-9V POST: number analyzed (Participants) | 214 | 112 | 1
  OPSONO-9V POST | 4693.7 [4099 to 5374.6] | 958.8 [680 to 1351.8] | 367 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-14 PRE: number analyzed (Participants) | 211 | 111 | 1
  OPSONO-14 PRE | 673.1 [573.1 to 790.6] | 826.7 [669.3 to 1021] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-14 POST: number analyzed (Participants) | 213 | 112 | 1
  OPSONO-14 POST | 6209 [5299.3 to 7274.8] | 819.1 [651.4 to 1030.1] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-18C PRE: number analyzed (Participants) | 207 | 112 | 1
  OPSONO-18C PRE | 26.3 [21.1 to 32.6] | 11.5 [8.2 to 16] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-18C POST: number analyzed (Participants) | 214 | 109 | 1
  OPSONO-18C POST | 2181 [1900.1 to 2503.4] | 12.7 [9.1 to 17.7] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-19F PRE: number analyzed (Participants) | 204 | 110 | 1
  OPSONO-19F PRE | 83.4 [64.7 to 107.6] | 21.1 [13.5 to 32.9] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-19F POST: number analyzed (Participants) | 212 | 108 | 1
  OPSONO-19F POST | 3496.3 [2938.8 to 4159.6] | 20.9 [13.7 to 31.8] | 191 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-23F PRE: number analyzed (Participants) | 209 | 111 | 1
  OPSONO-23F PRE | 600.5 [417.6 to 863.4] | 1048 [561.5 to 1956.1] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-23F POST: number analyzed (Participants) | 214 | 111 | 1
  OPSONO-23F POST | 7057.2 [5896.6 to 8446.1] | 1758.3 [949.4 to 3256.5] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)

5. Secondary Outcome: Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes 6A and 19A (Primary Immunization)
Description: Concentrations were given in microgram per millilitre (µg/mL) and were expressed in geometric mean antibody concentrations. Cross-reactive pneumococcal vaccine serotypes assessed were 6A and 19A. The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 µg/mL. Antibody concentrations < 0.05 µg/mL were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
Time Frame: 1 month following primary immunization (at Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 10Pn Group | DTPa Group
Number analyzed (Participants) | 231 | 121
μg/mL
  Anti-6A: number analyzed (Participants) | 230 | 121
  Anti-6A | 0.41 [0.34 to 0.49] | 0.04 [0.03 to 0.04]
  Anti-19A | 0.48 [0.4 to 0.57] | 0.04 [0.04 to 0.05]

6. Secondary Outcome: Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes 6A and 19A (Booster Immunization)
Description: Concentrations were given in microgram per millilitre (µg/mL) and were expressed in geometric mean antibody concentrations. Cross-reactive pneumococcal vaccine serotypes assessed were 6A and 19A. The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 µg/mL. Antibody concentrations < 0.05 g/mL were given an arbitrary value of half the cut-off for the purpose of GMC calculation. Administration of catch-up pneumococcal vaccination with a licensed product other than Synflorix was allowed in the DTPa Group at least 7 days before DTPa vaccine booster dose. Thus, for this booster phase analysis, the DTPa Group was further split in DTPa + Prevenar Group and DTPa - no Prevenar Group.
Time Frame: Prior to (PRE, at Month 14-16) and one month after booster (POST, at Month 15-17) immunization
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 10Pn Group | DTPa + Prevenar Group | DTPa - no Prevenar Group
Number analyzed (Participants) | 214 | 114 | 1
μg/mL
  Anti-6A PRE: number analyzed (Participants) | 209 | 114 | 1
  Anti-6A PRE | 0.61 [0.5 to 0.75] | 0.19 [0.14 to 0.26] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-6A POST | 2.72 [2.24 to 3.3] | 0.21 [0.16 to 0.27] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-19A PRE | 0.57 [0.45 to 0.71] | 0.12 [0.09 to 0.16] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  Anti-19A POST | 5.16 [4.18 to 6.37] | 0.15 [0.11 to 0.2] | 0.03 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)

7. Secondary Outcome: Opsonophagocytic Titers Against Cross-reactive Pneumococcal Serotypes 6A and 19A (Primary Immunization)
Description: Cross-reactive pneumococcal vaccine serotypes assessed were 6A and 19A and were calculated, expressed as geometric mean titers (GMTs). The seropositivity cut-off for the assay was ≥ 8. Antibody titers < 8 were given an arbitrary value of half the cut-off for the purpose of GMT calculation.
Time Frame: 1 month following primary immunization (at Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10Pn Group | DTPa Group
Number analyzed (Participants) | 213 | 115
Titers
  Opsono-6A: number analyzed (Participants) | 206 | 106
  Opsono-6A | 339.6 [253.8 to 454.4] | 4.6 [4.1 to 5.1]
  Opsono-19A | 34.3 [26.2 to 44.9] | 4.3 [4 to 4.6]

8. Secondary Outcome: Opsonophagocytic Titers Against Cross-reactive Pneumococcal Serotypes 6A and 19A (Booster Immunization)
Description: Cross-reactive pneumococcal vaccine serotypes assessed were 6A and 19A and were calculated, expressed as geometric mean titers (GMTs). The seropositivity cut-off for the assay was ≥ 8. Antibody titers < 8 were given an arbitrary value of half the cut-off for the purpose of GMT calculation. Administration of catch-up pneumococcal vaccination with a licensed product other than Synflorix was allowed in the DTPa Group at least 7 days before DTPa vaccine booster dose. Thus, for this booster phase analysis, the DTPa Group was further split in DTPa + Prevenar Group and DTPa - no Prevenar Group.
Time Frame: Prior to (PRE, at Month 14-16) and one month after booster (POST, at Month 15-17) immunization
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10Pn Group | DTPa + Prevenar Group | DTPa - no Prevenar Group
Number analyzed (Participants) | 213 | 111 | 1
Titers
  OPSONO-6A PRE: number analyzed (Participants) | 196 | 107 | 1
  OPSONO-6A PRE | 138.5 [103.3 to 185.7] | 60.4 [35.2 to 103.7] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-6A POST: number analyzed (Participants) | 212 | 107 | 1
  OPSONO-6A POST | 767.9 [593.1 to 994.1] | 103.3 [60.4 to 176.6] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-19A PRE | 13.1 [10.1 to 16.9] | 7.7 [5.5 to 10.6] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)
  OPSONO-19A POST: number analyzed (Participants) | 212 | 109 | 1
  OPSONO-19A POST | 431.4 [330.9 to 562.4] | 8.6 [6 to 12.2] | 4 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable because number of subjects with concentrations within the specified range = 0)

9. Secondary Outcome: Concentrations of Antibodies Against Protein D (PD) (Primary Immunization)
Description: Anti-protein D (Anti-PD) antibody concentrations by Enzyme-Linked Immunosorbent Assay (ELISA) were calculated, expressed as geometric mean concentrations (GMCs) in ELISA unit per milli-liter (EL.U/mL) and tabulated. The seropositivity cut-off for the assay was ≥ 100 EL.U/mL. Antibody concentrations < 100 EL.U/mL were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
Time Frame: 1 month following primary immunization (at Month 3)
Population: The analysis was performed on the ATP cohort for immunogenicity for primary epoch, which included all evaluable subjects for whom assay results were available for antibodies against Protein D after primary vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10Pn Group | DTPa Group
Number analyzed (Participants) | 229 | 119
EL.U/mL | 2548.6 [2315.1 to 2805.7] | 87.9 [75.8 to 102]

10. Secondary Outcome: Concentrations of Antibodies Against Protein D (PD) (Booster Immunization)
Description: as for outcome 9
Time Frame: Prior to (PRE, at Month 14-16) and one month after booster (POST, at Month 15-17) immunization
Population: Analysis was performed on the ATP cohort for immunogenicity for booster epoch, which included all evaluable subjects with assay results available for antibodies against Protein D before and after booster vaccination. Analysis was performed on the 10Pn Group and only on the pooled DTPa booster Group, i.e subjects with or without Prevenar vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Groups:
- DTPa Booster Group: Subjects from DTPa + Prevenar Group and DTPa - no Prevenar Group.
Arm/Group | 10Pn Group | DTPa Booster Group
Number analyzed (Participants) | 214 | 113
EL.U/mL
  Anti-PD PRE: number analyzed (Participants) | 210 | 112
  Anti-PD PRE | 702.6 [601 to 821.5] | 82.3 [71.7 to 94.5]
  Anti-PD POST | 2916.9 [2552.9 to 3332.7] | 86.9 [75.1 to 100.4]

11. Secondary Outcome: Concentrations of Antibodies Against Diphtheria Toxoid (DT) and Tetanus Toxoid (TT)(Primary Immunization)
Description: Concentrations of antibodies are presented as geometric mean concentrations expressed as International units per millilitre (IU/mL). Seroprotection status, defined as Anti-DT or Anti-TT antibody concentration equal to or greater than 0.1 IU/mL.
Time Frame: 1 month following primary immunization (at Month 3)
Population: The analysis was performed on the ATP cohort for immunogenicity for primary epoch, which included all evaluable subjects for whom assay results were available for antibodies against Diphtheria Toxoid or Tetanus Toxoid after primary vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 10Pn Group | DTPa Group
Number analyzed (Participants) | 230 | 120
IU/mL
  Anti-DT: number analyzed (Participants) | 229 | 120
  Anti-DT | 5.363 [5.002 to 5.749] | 3.829 [3.464 to 4.233]
  Anti-TT | 5.427 [4.94 to 5.962] | 3.626 [3.174 to 4.143]

12. Secondary Outcome: Concentrations of Antibodies Against Diphtheria Toxoid (DT) and Tetanus Toxoid (TT)(Booster Immunization)
Description: as for outcome 11
Time Frame: Prior to (PRE, at Month 14-16) and one month after booster (POST, at Month 15-17) immunization
Population: Analysis was performed on the ATP cohort for immunogenicity for booster epoch, which included all evaluable subjects with assay results available for antibodies against DT or TT before and after booster vaccination. Analysis was performed on the 10Pn Group and only on the pooled DTPa booster Group, i.e subjects with or without Prevenar vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 10Pn Group | DTPa Booster Group
Number analyzed (Participants) | 214 | 113
IU/mL
  Anti-DT PRE: number analyzed (Participants) | 211 | 112
  Anti-DT PRE | 0.615 [0.556 to 0.679] | 0.717 [0.618 to 0.833]
  Anti-DT POST | 15.977 [14.573 to 17.515] | 10.814 [9.684 to 12.075]
  Anti-TT PRE: number analyzed (Participants) | 210 | 113
  Anti-TT PRE | 2.043 [1.677 to 2.489] | 1.352 [1.038 to 1.762]
  Anti-TT POST | 11.057 [9.949 to 12.287] | 6.278 [5.334 to 7.389]

13. Secondary Outcome: Concentrations of Antibodies Against Pertussis (PT) and Filamentous Haemagglutinin (FHA)(Primary Immunization)
Description: Concentrations of antibodies are presented as geometric mean concentrations expressed as Enzyme-Linked Immuno-Sorbent Assay (ELISA) units per millilitre (EL.U/mL). Seropositivity was defined as an antibody concentration equal to or greater than 5 EL.U/mL
Time Frame: 1 month following primary immunization (at Month 3)
Population: The analysis was performed on the ATP cohort for immunogenicity for primary epoch, which included all evaluable subjects for whom assay results were available for antibodies against Pertussis or Filamentous haemagglutinin after primary vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10Pn Group | DTPa Group
Number analyzed (Participants) | 231 | 121
EL.U/mL
  Anti-PT | 123.2 [115.2 to 131.7] | 133.1 [119.5 to 148.3]
  Anti-FHA | 308.6 [284.8 to 334.3] | 365 [327.9 to 406.2]

14. Secondary Outcome: Concentrations of Antibodies Against Pertussis (PT) and Filamentous Haemagglutinin (FHA)(Booster Immunization)
Description: as for outcome 13
Time Frame: Prior to (PRE, at Month 14-16) and one month after booster (POST, at Month 15-17) immunization
Population: Analysis was performed on the ATPcohort for immunogenicity for booster epoch, which included all evaluable subjects with assay results available for antibodies against PT or FHA before and after booster vaccination. Analysis was performed on the 10Pn Group and only on the pooled DTPa booster Group, i.e. subjects with or without Prevenar vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10Pn Group | DTPa Booster Group
Number analyzed (Participants) | 214 | 114
EL.U/mL
  Anti-PT PRE: number analyzed (Participants) | 210 | 113
  Anti-PT PRE | 14.9 [13.2 to 16.8] | 18.1 [15.1 to 21.7]
  Anti-PT POST: number analyzed (Participants) | 213 | 114
  Anti-PT POST | 158.4 [143.7 to 174.7] | 204 [176.7 to 235.6]
  Anti-FHA PRE: number analyzed (Participants) | 210 | 114
  Anti-FHA PRE | 37.9 [33.3 to 43.1] | 48.4 [40.6 to 57.8]
  Anti-FHA POST | 460.6 [421.2 to 503.7] | 584.5 [512.6 to 666.6]

15. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms After Primary Vaccination
Description: Solicited local AEs assessed were pain, redness and swelling. Any = incidence of any local symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling above 30 millimetre.
Time Frame: During the 8-day (Days 0-7) after each primary vaccine dose
Population: The analysis was performed on the Total Vaccinated cohort for primary epoch, which included all subjects having received at least one of the 3 primary vaccination doses and who had their symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn Group | DTPa Group
Number analyzed (Participants) | 237 | 123
Participants
  Any pain Dose 1 | 83 | 19
  Grade 3 pain Dose 1 | 1 | 0
  Any redness Dose 1 | 182 | 71
  Grade 3 Redness Dose 1 | 10 | 0
  Any swelling Dose 1 | 126 | 33
  Grade 3 Swelling Dose 1 | 16 | 0
  Any pain Dose 2: number analyzed (Participants) | 235 | 123
  Any pain Dose 2 | 74 | 26
  Grade 3 pain Dose 2: number analyzed (Participants) | 235 | 123
  Grade 3 pain Dose 2 | 0 | 0
  Any redness Dose 2: number analyzed (Participants) | 235 | 123
  Any redness Dose 2 | 200 | 96
  Grade 3 Redness Dose 2: number analyzed (Participants) | 235 | 123
  Grade 3 Redness Dose 2 | 25 | 4
  Any swelling Dose 2: number analyzed (Participants) | 235 | 123
  Any swelling Dose 2 | 160 | 75
  Grade 3 Swelling Dose 2: number analyzed (Participants) | 235 | 123
  Grade 3 Swelling Dose 2 | 26 | 4
  Any pain Dose 3: number analyzed (Participants) | 233 | 122
  Any pain Dose 3 | 63 | 23
  Grade 3 pain Dose 3: number analyzed (Participants) | 233 | 122
  Grade 3 pain Dose 3 | 1 | 0
  Any redness Dose 3: number analyzed (Participants) | 233 | 122
  Any redness Dose 3 | 178 | 84
  Grade 3 Redness Dose 3: number analyzed (Participants) | 233 | 122
  Grade 3 Redness Dose 3 | 24 | 0
  Any swelling Dose 3: number analyzed (Participants) | 233 | 122
  Any swelling Dose 3 | 142 | 65
  Grade 3 Swelling Dose 3: number analyzed (Participants) | 233 | 122
  Grade 3 Swelling Dose 3 | 27 | 1

16. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms After Booster Vaccination
Description: as for outcome 15
Time Frame: During the 8-day (Days 0-7) period following booster vaccination
Population: The analysis was performed on the Total Vaccinated cohort for booster epoch, which included all subjects having received the booster dose and who had their symptoms sheet filled in. Analysis was performed on the 10Pn Group and only on the pooled DTPa booster Group, i.e subjects with or without Prevenar vaccination.
Measure: Number; unit: Subjects
Arm/Group | 10Pn Group | DTPa Booster Group
Number analyzed (Participants) | 228 | 120
Subjects
  Any pain | 134 | 47
  Grade 3 pain | 12 | 0
  Any redness | 197 | 102
  Redness > 30 mm | 72 | 20
  Any swelling | 180 | 90
  Swelling > 30 mm | 65 | 18

17. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms After Primary Vaccination
Description: General AEs = drowsiness, fever (axillary ≥ 37.5 degrees Celsius), irritabilityand loss of appetite, vomiting. Any= Incidence of any symptom regardless of intensity grade or relationship to vaccination. Grade 3 drowsiness = prevented normal activity. Grade 3 irritability = crying that could not be comforted/ prevented normal activity. Grade 3 loss of appetite = not eating at all. Grade 3 fever = > 39.5°C Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 8-day (Days 0-7) after each primary vaccine dose
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn Group | DTPa Group
Number analyzed (Participants) | 237 | 123
Participants
  Any drowsiness Dose 1 | 67 | 24
  Grade 3 drowsiness Dose 1 | 3 | 0
  Related drowsiness Dose 1 | 24 | 6
  Any Fever Dose 1 | 61 | 20
  Grade 3 Fever Dose 1 | 1 | 0
  Related fever Dose 1 | 20 | 5
  Any irritability Dose 1 | 100 | 43
  Grade 3 irritability Dose 1 | 6 | 3
  Related irritability Dose 1 | 40 | 12
  Any loss of appetite Dose 1 | 32 | 12
  Grade 3 loss of appetite Dose 1 | 0 | 0
  Related loss of appetite Dose 1 | 4 | 1
  Any drowsiness Dose 2: number analyzed (Participants) | 235 | 123
  Any drowsiness Dose 2 | 67 | 34
  Grade 3 drowsiness Dose 2: number analyzed (Participants) | 235 | 123
  Grade 3 drowsiness Dose 2 | 2 | 0
  Related drowsiness Dose 2: number analyzed (Participants) | 235 | 123
  Related drowsiness Dose 2 | 26 | 9
  Any Fever Dose 2: number analyzed (Participants) | 235 | 123
  Any Fever Dose 2 | 65 | 22
  Grade 3 Fever Dose 2: number analyzed (Participants) | 235 | 123
  Grade 3 Fever Dose 2 | 0 | 0
  Related fever Dose 2: number analyzed (Participants) | 235 | 123
  Related fever Dose 2 | 31 | 7
  Any irritability Dose 2: number analyzed (Participants) | 235 | 123
  Any irritability Dose 2 | 88 | 45
  Grade 3 irritability Dose 2: number analyzed (Participants) | 235 | 123
  Grade 3 irritability Dose 2 | 4 | 0
  Related irritability Dose 2: number analyzed (Participants) | 235 | 123
  Related irritability Dose 2 | 30 | 12
  Any loss of appetite Dose 2: number analyzed (Participants) | 235 | 123
  Any loss of appetite Dose 2 | 27 | 7
  Grade 3 loss of appetite Dose 2: number analyzed (Participants) | 235 | 123
  Grade 3 loss of appetite Dose 2 | 0 | 0
  Related loss of appetite Dose 2: number analyzed (Participants) | 235 | 123
  Related loss of appetite Dose 2 | 7 | 2
  Any drowsiness Dose 3: number analyzed (Participants) | 233 | 122
  Any drowsiness Dose 3 | 41 | 25
  Grade 3 drowsiness Dose 3: number analyzed (Participants) | 233 | 122
  Grade 3 drowsiness Dose 3 | 0 | 0
  Related drowsiness Dose 3: number analyzed (Participants) | 233 | 122
  Related drowsiness Dose 3 | 15 | 10
  Any Fever Dose 3: number analyzed (Participants) | 233 | 122
  Any Fever Dose 3 | 51 | 21
  Grade 3 Fever Dose 3: number analyzed (Participants) | 233 | 122
  Grade 3 Fever Dose 3 | 2 | 0
  Related fever Dose 3: number analyzed (Participants) | 233 | 122
  Related fever Dose 3 | 21 | 2
  Any irritability Dose 3: number analyzed (Participants) | 233 | 122
  Any irritability Dose 3 | 80 | 31
  Grade 3 irritability Dose 3: number analyzed (Participants) | 233 | 122
  Grade 3 irritability Dose 3 | 3 | 0
  Related irritability Dose 3: number analyzed (Participants) | 233 | 122
  Related irritability Dose 3 | 31 | 10
  Any loss of appetite Dose 3: number analyzed (Participants) | 233 | 122
  Any loss of appetite Dose 3 | 25 | 7
  Grade 3 loss of appetite Dose 3: number analyzed (Participants) | 233 | 122
  Grade 3 loss of appetite Dose 3 | 0 | 0
  Related loss of appetite Dose 3: number analyzed (Participants) | 233 | 122
  Related loss of appetite Dose 3 | 5 | 0

18. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms After Booster Vaccination
Description: Solicited general AEs = drowsiness, irritability, loss of appetite and fever (axillary ≥ 37.5 degrees Celsius). Any= Incidence of any symptom regardless of intensity grade or relationship to vaccination. Grade 3: drowsiness = prevented normal activity. irritability = crying that could not be comforted/ prevented normal activity. loss of appetite = not eating at all. Fever = temperature > 39.5°C Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 8-day (Days 0-7) period following booster vaccination
Population: as for outcome 16
Measure: Number; unit: Subjects
Arm/Group | 10Pn Group | DTPa Booster Group
Number analyzed (Participants) | 228 | 120
Subjects
  Any drowsiness | 69 | 30
  Grade 3 drowsiness | 3 | 3
  Related drowsiness | 19 | 7
  Fever >= 37.5°C | 90 | 24
  Fever > 39.5°C | 6 | 0
  Related fever | 41 | 11
  Any irritability | 90 | 35
  Grade 3 irritability | 8 | 2
  Related irritability | 36 | 10
  Any loss of appetite | 48 | 17
  Grade 3 loss of appetite | 4 | 1
  Related loss of appetite | 12 | 2

19. Secondary Outcome: Number of Subjects With Unsolicited AEs After Primary Vaccination
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within the 31-day (Days 0-30) post-primary vaccination period, across doses
Population: The analysis was performed on the Total Vaccinated cohort for primary epoch, which included all subjects having received at least one of the 3 primary vaccination doses.
Measure: Number; unit: Subjects
Arm/Group | 10Pn Group | DTPa Group
Number analyzed (Participants) | 237 | 123
Subjects | 193 | 97

20. Secondary Outcome: Number of Subjects With Unsolicited AEs After Booster Vaccination
Description: as for outcome 19
Time Frame: Within the 31-day (Days 0-30) post booster vaccination period
Population: The analysis was performed on the Total Vaccinated cohort for booster epoch, which included all subjects having received the booster dose. Analysis was performed on the 10Pn Group and only on the pooled DTPa booster Group, i.e subjects with or without Prevenar vaccination.
Measure: Number; unit: Subjects
Arm/Group | 10Pn Group | DTPa Booster Group
Number analyzed (Participants) | 228 | 120
Subjects | 132 | 66

21. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: From study start at Month 0 up to study end at Month 15-17
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn Group | DTPa Group
Number analyzed (Participants) | 237 | 123
Participants | 28 | 19

ADVERSE EVENTS:
Time Frame: Solicited AEs: within 8 days (Day 0 - Day 7) after any vaccine dose; Unsolicited AEs: within 31 days (Day 0 - Day 30) after any vaccine dose. SAEs: from Dose 1 up to Study End (Day 0 to Month 15-17)
Description: All-causes mortality, SAEs and other AEs collection was made for primary vaccination phase groups, including all vaccinated subjects in the study.
Arm/Group | 10Pn Group | DTPa Group
All-Cause Mortality (participants affected / at risk) | 1/237 | 0/123
Serious Adverse Events (participants affected / at risk) | 28/237 | 19/123
Other Adverse Events (participants affected / at risk) | 236/237 | 122/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10Pn Group (N=237) | DTPa Group (N=123)
Ear malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Faciodigitogenital dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Strabismus (Eye disorders) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Sudden infant death syndrome (General disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Acute tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 3 (4) | 3 (3)
Bronchopneumonia (Infections and infestations) | 1 (1) | 1 (1)
Croup infectious (Infections and infestations) | 0 (0) | 3 (3)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (4) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (2)
Meningitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 6 (7) | 1 (1)
Pneumonia adenoviral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 5 (5) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (2) | 0 (0)
Febrile convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Myelitis transverse (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Fibrinous bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tuberculid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Kawasaki's disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10Pn Group (N=237) | DTPa Group (N=123)
Bronchitis (Infections and infestations) | 17 (21) | 15 (18)
Conjunctivitis (Eye disorders) | 18 (22) | 9 (13)
Decreased appetite (Metabolism and nutrition disorders) | 91 (133) | 37 (43)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 15 (19) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 29 (32) | 14 (14)
Eczema (Skin and subcutaneous tissue disorders) | 49 (65) | 25 (28)
Erythema (Skin and subcutaneous tissue disorders) | 230 (768) | 114 (368)
Gastroenteritis (Infections and infestations) | 18 (19) | 5 (5)
Impetigo (Infections and infestations) | 5 (5) | 8 (9)
Injection site induration (General disorders) | 56 (86) | 23 (34)
Irritability (Psychiatric disorders) | 177 (358) | 81 (154)
Nasopharyngitis (Infections and infestations) | 41 (60) | 24 (41)
Otitis media (Infections and infestations) | 9 (10) | 7 (7)
Pain (General disorders) | 167 (354) | 62 (115)
Pyrexia (General disorders) | 156 (284) | 64 (92)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 4 (4)
Somnolence (Nervous system disorders) | 131 (244) | 63 (113)
Swelling (General disorders) | 214 (610) | 113 (265)
Upper respiratory tract infection (Infections and infestations) | 85 (131) | 43 (69)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.